CLINICAL TRIAL: NCT04356625
Title: Maximum Expiratory Pressure in Induced Cough as a Predictor of Extubation Failure in Intensive Care Unit Patients on Mechanical Ventilation Ready to Extubate. A Single-arm Open Clinical Trial.
Brief Title: Maximum Expiratory Pressure in Induced Cough as a Predictor of Extubation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Nacional Profesor Alejandro Posadas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 209LUP0S0/18
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Airway Extubation
Keywords: airway extubation; maximal expiratory pressure; induced cough; ventilator weaning

STUDY DESIGN:
Intervention Model Description: Single-arm clinical trial to establish diagnostic performance of MEPic
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MEPic (Other): * Ready for extubation (pass SBT)
  * Measurement of maximum expiratory pressure during the induced cough (MEPic)
  Interventions: Diagnostic Test: MEPic

INTERVENTIONS:
Diagnostic Test: MEPic — * patient in the supine position sitting 45° to 60°,
  * closed suction catheter was removed
  * a 90° elbow was placed and a bacterial filter in series with endotracheal tube
  * adapter was also coupled to the aneroid pressure gauge
  * in series an inspiratory unidirectional valve was placed that did not allow expiration
  * 2 ml of physiological solution was slowly instilled through the port in the 90º elbow to cause induced cough

SUMMARY:
Clinical trial for the evaluation of diagnostic tests. The sample was composed of adults under mechanical ventilation who passed the spontaneous breathing trial and was ready to be extubated. The maximum expiratory pressure measured in the usual way and the maximum expiratory pressure generated during the induced cough were taken as predictor variables. The outcome variable was extubation failure, measured at 72 hours and at 7 days.

DETAILED DESCRIPTION:
After completing the spontaneous breathing trial (SBT), with the extubation decision defined by the physician in charge of the patient and maximal expiratory pressure (MEP) as usually measured greater than 30 centimeters of water (cmH2O). Following this, the patient was allowed to rest for 5 minutes in the same condition. With the patient in the supine position sitting 45 ° to 60 °, the closed suction catheter was removed, an elbow was placed at 90 ° and a bacterial filter in series with the endotracheal tube (ET), an adapter was also coupled with a outlet port to the aneroid pressure gauge. In series an inspiratory unidirectional valve was placed that did not allow expiration. Immediately 2 ml of physiological solution was slowly instilled through the port in the 90º elbow to trigger the cough reflex. The presence or absence of reflex cough and the MEP during induced cough (MEPic) value were verified.

As a safety method, the procedures were stopped if the patient presented signs of intolerance such as respiratory rate (RF)> 35 breaths per minute, saturation <90%, heart rate (HR)> 140 beats per minute or increase of 20 % of resting levels.

ELIGIBILITY:
Inclusion Criteria:

* Under mechanical ventilation via endotracheal tube in a period greater than 48 hours
* Passing the spontaneous breathing trial an be ready for extubation.
* Agree to participate in the study and sign the informed consent by the patient or family member

Exclusion Criteria:

* tracheostomized prior to admission to mechanical ventilation
* history of neuromuscular disease
* presence of unstable heart disease
* received upper digestive surgery
* presence of uncontained enterocutaneous fistula
* candidates for non-invasive ventilation as a modality of interface exchange for extubation or as a preventive modality
* patients who did not reach a MEP (habitual) of 30 cmH20 since they are not extubated by the extubation protocol of our institution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
Extubation failure | 72 hours
  Endotracheal tube removal failure
Extubation failure | 7 days
  Endotracheal tube removal failure

CONTACTS AND LOCATIONS:
Overall Officials: Ladislao P Diaz-Ballve, Lic., Principal Investigator — Hospital Nacional Profesor Alejandro Posadas
Locations (1):
- Ladislao Diaz Ballve, Haedo, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrera M, Urrutia JG, Ardariz CB, Porra ML, Gamarra C, Ballve LPD. Maximal expiratory pressure compared with maximal expiratory pressure during induced cough as a predictor of extubation failure. Crit Care Sci. 2023 Mar 1;35(1):37-43. doi: 10.5935/2965-2774.20230275-en. PMID 37712728